CLINICAL TRIAL: NCT02492165
Title: Immunogenicity and Safety of a Single Primary Dose of a Live Attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®) Given to Healthy Subjects in Vietnam
Brief Title: Study of a Single Primary Dose Live Attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®) in Healthy Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JEC13; U1111-1143-8142 (Other: WHO); NCT02821221 (obsolete NCT alias)
Record Dates: First submitted 2015-07-05; First posted 2015-07-08 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Japanese Encephalitis
Keywords: Japanese Encephalitis; Japanese encephalitis chimeric virus vaccine; IMOJEV®; Live attenuated vaccine
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Age 9 Months through 4 Years Group (Experimental): Participants age 9 Months through 4 Years old at enrollment
  Interventions: Biological: Live attenuated Japanese encephalitis chimeric virus vaccine (IMOJEV®)
- Age 5 Years through 11 Years Group (Experimental): Participants age 5 Years through 11 Years old at enrollment
  Interventions: Biological: Live attenuated Japanese encephalitis chimeric virus vaccine (IMOJEV®)
- Age 12 Years through 17 Years Group (Experimental): Participants age 12 Years through 17 Years old at enrollment
  Interventions: Biological: Live attenuated Japanese encephalitis chimeric virus vaccine (IMOJEV®)
- Age 18 Years through 60 Years Group (Experimental): Participants age 18 Years through 60 Years old at enrollment
  Interventions: Biological: Live attenuated Japanese encephalitis chimeric virus vaccine (IMOJEV®)

INTERVENTIONS:
Biological: Live attenuated Japanese encephalitis chimeric virus vaccine (IMOJEV®) — 0.5 mL, Subcutaneous
  Other Names: IMOJEV®
  Arms: Age 9 Months through 4 Years Group
Biological: Live attenuated Japanese encephalitis chimeric virus vaccine (IMOJEV®) — 0.5 mL, Subcutaneous
  Other Names: IMOJEV®
  Arms: Age 5 Years through 11 Years Group
Biological: Live attenuated Japanese encephalitis chimeric virus vaccine (IMOJEV®) — 0.5 mL, Subcutaneous
  Other Names: IMOJEV®
  Arms: Age 12 Years through 17 Years Group
Biological: Live attenuated Japanese encephalitis chimeric virus vaccine (IMOJEV®) — 0.5 mL, Subcutaneous
  Other Names: IMOJEV®
  Arms: Age 18 Years through 60 Years Group

SUMMARY:
The purpose of this study is to describe the immunogenicity and safety of IMOJEV® in adult and pediatric populations in Vietnam and serve a bridging study to compare immunogenicity, reactogenicity, and safety data obtained with IMOJEV® in the Vietnamese population with data from other Asian pediatric populations.

Primary objective:

- To describe the safety profile of a single dose of IMOJEV®.

Secondary objectives:

* To evaluate the immune response to JE 28 days after the administration of a single dose of IMOJEV® in healthy Vietnamese subjects aged from 9 months to 60 years.

DETAILED DESCRIPTION:
Study participants will be enrolled by age group and will each receive one injection of IMOJEV® on Day 0 given as primary vaccination. They will be assessed for immunogenicity and safety, post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 9 months through 60 years on the day of inclusion.
* For adults: Informed consent form has been signed and dated by the subject. For minors: Informed consent form has been signed and dated by the parent or legally acceptable representative. In addition, in accordance with the Institution Ethics Committee / Institution Review Board requirements and as appropriate for the age of the subject, the subject may be required to sign and date the informed consent form if aged 12 to 17 years or assent form if aged 8 to 11 years.
* Subject and parent(s)/legally acceptable representative(s) are able to attend all scheduled visits and comply with all study procedures.

Exclusion Criteria:

* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche, or post-menopausal for at least 1 year, or surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination).
* Participation at the time of study enrollment (or in the 4 weeks preceding the study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or a medical procedure.
* Receipt of any vaccine in the 4 weeks preceding the study vaccination or planned receipt of any vaccine in the 4 weeks following the study vaccination, except for inactivated influenza vaccination, which may be received at least 2 weeks before the study vaccine
* Previous vaccination against flavivirus disease, including Japanese Encephalitis (JE), dengue, and yellow fever.
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months that might interfere with the assessment of the immune response.
* Known or suspected congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy (for more than 2 consecutive weeks within the 4 weeks preceding vaccination).
* History of flavivirus infection (confirmed either clinically, serologically, or virologically).
* History of central nervous system disorder or disease, including seizures.
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the study or to a vaccine containing any of the same substances.
* Known thrombocytopenia, contraindicating vaccination.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion.
* Febrile illness (temperature ≥ 38.0°C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment. A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided.
* Receipt of any chronic anti-viral in the 2 months preceding the study vaccination or planned receipt of any anti-viral in the 4 weeks following the study vaccination. Short-term antiviral drugs for flu or herpes can be administered provided there is a wash-out period of 1 week before the administration of the vaccine.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Ages: 9 Months to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 250 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- Preventive Medicine Centre of Hoa Binh Province, Hòa Bình, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Vu TD, Nguyen QD, Tran HTA, Bosch-Castells V, Zocchetti C, Houillon G. Immunogenicity and safety of a single dose of a live attenuated Japanese encephalitis chimeric virus vaccine in Vietnam: A single-arm, single-center study. Int J Infect Dis. 2018 Jan;66:137-142. doi: 10.1016/j.ijid.2017.10.010. Epub 2017 Nov 27. PMID 29081368
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 27 June 2015 to 24 August 2015 at 1 clinic center in Vietnam.
Pre-assignment Details: A total of 250 participants who met all inclusion and no exclusion criteria were enrolled and vaccinated.
Groups:
- 9 Months to 4 Years: Healthy participants aged 9 months to 4 years who received a single primary dose of a live attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®).
- 5 to 11 Years: Healthy participants aged 5 to 11 years who received a single primary dose of a live attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®).
- 12 to 17 Years: Healthy participants aged 12 to 17 years who received a single primary dose of a live attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®).
- 18 to 60 Years: Healthy participants aged 18 to 60 years who received a single primary dose of a live attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®).
Period: Overall Study
Arm/Group | 9 Months to 4 Years | 5 to 11 Years | 12 to 17 Years | 18 to 60 Years
Started | 100 | 60 | 60 | 30
Completed | 100 | 59 | 60 | 30
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 9 Months to 4 Years | 5 to 11 Years | 12 to 17 Years | 18 to 60 Years | Total
Number analyzed (Participants) | 100 | 60 | 60 | 30 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100 | 60 | 60 | 0 | 220
  Between 18 and 65 years | 0 | 0 | 0 | 30 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 0.7 (0.6) | 8.7 (1.5) | 13.9 (1.4) | 38.7 (10.0) | 15.75 (3.375)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 31 | 42 | 22 | 141
  Male | 54 | 29 | 18 | 8 | 109
Region of Enrollment [Number; unit: Participants]
  Vietnam | 100 | 60 | 60 | 30 | 250

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Injection Site Reactions and Systemic Events Following a Single Primary Dose of a Live Attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
Description: Solicited injection-site: ≤ 23 months age: Tenderness, Erythema, and Swelling. For ≥ 2 years age: Pain, Erythema, and Swelling. Solicited systemic reactions: ≤ 23 months age, Fever (temperature) Vomiting, Crying abnormal, Drowsiness, Appetite loss, Irritability, For ≥ 2 years age, Fever (temperature) Headache, Malaise, and Myalgia.
  Grade 3: Tenderness, Cries when injected limb is moved; Pain, Incapacitating, unable to perform usual activities or Significant; prevents daily activity (≥ 12 years); Erythema and Swelling (≤23 months to 11 years), ≥50 mm or >100 mm (≥ 12 years).
  Grade 3 Fever, > 39.5°C (≤ 23 months) or ≥39.0°C (≥ 2 years); Vomiting, ≥ 6 episodes per 24 hours; Crying abnormal, > 3 hours; Drowsiness, Sleeping most of the time; Appetite loss, Refuses ≥ 3 feeds / meals; Irritability, Inconsolable. Headache, Malaise, and Myalgia, Significant; prevents daily activity.
Time Frame: Day 0 up to Day 14 post-vaccination
Population: Solicited injection site and solicited systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | 9 Months to 4 Years | 5 to 11 Years | 12 to 17 Years | 18 to 60 Years
Number analyzed (Participants) | 100 | 60 | 60 | 30
Participants
  Injection-site Tenderness/Pain | 35 | 8 | 11 | 8
  Grade 3 Injection-site Tenderness/Pain | 0 | 0 | 0 | 0
  Injection-site Erythema | 6 | 3 | 0 | 0
  Grade 3 Injection-site Erythema | 0 | 0 | 0 | 0
  Injection-site Swelling | 1 | 1 | 0 | 0
  Grade 3 Injection-site Swelling | 0 | 0 | 0 | 0
  Fever | 14 | 0 | 0 | 0
  Grade 3 Fever | 2 | 1 | 0 | 0
  Vomiting | 12 | NA — Event was not solicited for this group | NA — Event was not solicited for this group | NA — Event was not solicited for this group
  Grade 3 Vomiting | 0 | NA — Event was not solicited for this group | NA — Event was not solicited for this group | NA — Event was not solicited for this group
  Crying abnormal | 20 | NA — Event was not solicited for this group | NA — Event was not solicited for this group | NA — Event was not solicited for this group
  Grade 3 Crying abnormal | 0 | NA — Event was not solicited for this group | NA — Event was not solicited for this group | NA — Event was not solicited for this group
  Drowsiness | 12 | NA — Event was not solicited for this group | NA — Event was not solicited for this group | NA — Event was not solicited for this group
  Grade 3 Drowsiness | 0 | NA — Event was not solicited for this group | NA — Event was not solicited for this group | NA — Event was not solicited for this group
  Appetite loss | 38 | NA — Event was not solicited for this group | NA — Event was not solicited for this group | NA — Event was not solicited for this group
  Grade 3 Appetite loss | 1 | NA — Event was not solicited for this group | NA — Event was not solicited for this group | NA — Event was not solicited for this group
  Irritability | 21 | NA — Event was not solicited for this group | NA — Event was not solicited for this group | NA — Event was not solicited for this group
  Grade 3 Irritability | 0 | NA — Event was not solicited for this group | NA — Event was not solicited for this group | NA — Event was not solicited for this group
  Headache | NA — Event was not solicited for this group | 9 | 14 | 10
  Grade 3 Headache | NA — Event was not solicited for this group | 0 | 0 | 0
  Malaise | 1 | 8 | 16 | 9
  Grade 3 Malaise | 0 | 0 | 0 | 0
  Myalgia | 0 | 5 | 9 | 5
  Grade 3 Myalgia | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With Japanese Encephalitis Seroprotection Following a Single Primary Dose of a Live Attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
Description: Neutralizing antibodies were measured using a Japanese encephalitis chimeric virus (JE CV) 50% plaque reduction neutralization test (PRNT50). Seroprotection was defined as antibody titer levels ≥10 (1/dil).
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Seroprotection was assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | 9 Months to 4 Years | 5 to 11 Years | 12 to 17 Years | 18 to 60 Years
Number analyzed (Participants) | 76 | 60 | 19 | 5
Percentage of participants
  Pre-vaccination (Day 0) | 0.0 | 0.0 | 0.0 | 0.0
  Post-vaccination (Day 28) | 97.4 | 100.0 | 100.0 | 100.0

3. Primary Outcome: Percentage of Participants With Japanese Encephalitis Seroconversion Following a Single Primary Dose of a Live Attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
Description: Neutralizing antibodies were measured using a Japanese encephalitis chimeric virus (JE CV) 50% plaque reduction neutralization test (PRNT50). Seroconversion was defined as participants with a pre-vaccination titer <10 (1/dil) and post-vaccination titer ≥10 (1/dil) or participants with pre vaccination titer ≥10 (1/dil) and a ≥4-fold increase from pre- to post-vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Seroconversion was assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | 9 Months to 4 Years | 5 to 11 Years | 12 to 17 Years | 18 to 60 Years
Number analyzed (Participants) | 76 | 60 | 19 | 5
Percentage of participants | 97.4 | 100.0 | 100.0 | 100.0

4. Primary Outcome: Summary of Geometric Mean Titers of Japanese Encephalitis Antibodies Following a Single Primary Dose of a Live Attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®)
Description: Neutralizing antibodies were measured using a Japanese encephalitis chimeric virus (JE CV) 50% plaque reduction neutralization test (PRNT50).
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric mean titers were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dil)
Arm/Group | 9 Months to 4 Years | 5 to 11 Years | 12 to 17 Years | 18 to 60 Years
Number analyzed (Participants) | 76 | 34 | 19 | 5
Titers (1/dil)
  Pre-vaccination (Day 0) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Post-vaccination (Day 28) | 277 [192 to 399] | 1738 [1055 to 2862] | 1481 [762 to 2878] | 970 [65.6 to 14352]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 up to Day 28 post vaccination.
Arm/Group | 9 Months to 4 Years | 5 to 11 Years | 12 to 17 Years | 18 to 60 Years
Serious Adverse Events (participants affected / at risk) | 1/100 | 0/60 | 1/60 | 0/30
Other Adverse Events (participants affected / at risk) | 38/100 | 9/60 | 16/60 | 10/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 9 Months to 4 Years (N=100) | 5 to 11 Years (N=60) | 12 to 17 Years (N=60) | 18 to 60 Years (N=30)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 9 Months to 4 Years (N=100) | 5 to 11 Years (N=60) | 12 to 17 Years (N=60) | 18 to 60 Years (N=30)
Diarrhea (Gastrointestinal disorders) | 5 (7) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Injection site Tenderness/Pain (General disorders) | 34 (34) | 8 (8) | 11 (11) | 8 (8)
Injection site Erythema (General disorders) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
Fever (General disorders) | 14 (14) | 7 (7) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 12 (12) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Crying abnormal (Psychiatric disorders) | 20 (20) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Drowsiness (Nervous system disorders) | 12 (12) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Appetite loss (Metabolism and nutrition disorders) | 38 (38) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Irritability (Psychiatric disorders) | 21 (21) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Headache (Nervous system disorders) | 0 (0) | 9 (9) | 14 (14) | 10 (10)
Malaise (General disorders) | 0 (0) | 8 (8) | 16 (16) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 9 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.